CLINICAL TRIAL: NCT02781506
Title: Phase II Trial of Nivolumab and Stereotactic Ablative Radiation Therapy (SAbR) for Metastatic Clear Cell Renal Cell Carcinoma (mRCC)
Brief Title: Nivolumab and Stereotactic Ablative Radiation Therapy (SAbR) for Metastatic Clear Cell Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Since the treatment landscape for metastatic kidney cancer changed, patients were not becoming eligible for this trial and therefore, the trial was terminated.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Raquibul Hannan, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 122015-052
Record Dates: First submitted 2016-05-19; First posted 2016-05-24 (Estimated); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab and SABR (Experimental): Nivolumab alone: IV, administered per standard of care according to institutional guidelines at the discretion of the treating medical oncologist, until disease progression or unacceptable toxicity. SABR, dose variable, in 1-3 fractions.
  Interventions: Drug: Nivolumab; Radiation: SAbR

INTERVENTIONS:
Drug: Nivolumab — Nivolumab IV, administered per standard of care according to institutional guidelines at the discretion of the treating medical oncologist
  Other Names: Opdivo
Radiation: SAbR — SAbR (1-3 lesions)
  Other Names: SBRT; Stereotactic Ablative Radiation Therapy

SUMMARY:
Nivolumab (brand name Opdivo): IV, administered per standard of care according to institutional guidelines at the discretion of the treating medical oncologist, until disease progression or unacceptable toxicity; SABR, dose variable, in 1-3 fractions.

DETAILED DESCRIPTION:
A single institution, safety lead-in phase II trial with SAbR to multiple metastatic sites concurrently administered with Nivolumab for patients with metastatic clear cell renal cell cancer who have failed at least one anti-angiogenic therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Willing and able to provide consent
* Pathologic diagnosis of metastatic RCC with clear cell component
* Measurable disease in at least 2 non-radiated sites. Progression or intolerance to at least one prior systemic anti-angiogenic therapy.
* Eligible for extra-CNS SAbR to 1-6 sites of disease
* Must have received at least one prior anti-angiogenic therapy in the advanced or metastatic setting. Prior cytokine therapy (eg, IL-2, IFN-α), vaccine therapy, or treatment with cytotoxic therapy is also allowed but not any other drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Previous treatment with surgery, radiation, chemotherapy, targeted agents (see above) are allowed provided that: Chemotherapy/Major surgery was administered > 14 days before the start Nivolumab; Minor surgery, radiation, or any targeted agents were administered > 7 days before the start of Nivolumab
* Performance status ECOG 0, 1, 2 or 3.
* Adequate organ and marrow function as defined below (obtained within 14 days of first dose of drug):

  * leukocytes≥ 2,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 50,000/mcl
  * total bilirubin ≤ 2mg/dL
  * AST(SGOT)/ALT(SPGT) ≤ 3 X institutional upper limit of normal
* Women of child-bearing potential

  * female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
  * must have a negative serum or urine pregnancy test within 24 hours prior to the start of investigational product.
  * Women must not be breastfeeding.
  * must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and contraception should be continued for a period of 30 days plus the time required for the investigational drug to undergo five half lives.
  * Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
  * Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Contraception should be continued for a period of 90 days plus the time required for the investigational drug to undergo five half lives. This is equivalent to 31 weeks after discontinuation of Nivolumab.
* Adequate Renal function with Cr ≤ 2.5 mg/dL.

Exclusion Criteria:

* Subjects who have had major surgery (such as nephrectomy) or chemotherapy within 2 weeks prior to first dose of drug
* Subjects who have had radiation therapy within 2 weeks prior to first dose of drug
* Uncontrolled adrenal insufficiency or active chronic liver disease
* Any history of CNS metastases that is not adequately treated with surgery or SABR >14 days prior.
* Prior treatment with any anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Any positive history for HIV/AIDS, HTLV, hepatitis B or hepatitis C virus indicating acute or chronic infection.
* Any active known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose of study drug. Inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalent are permitted (although not encouraged) in the absence of active autoimmune disease.
* Subjects with life expectancy < 6 months
* Subjects receiving any other investigational or standard antineoplastic agents.
* Prior malignancies active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, breast?, or etc.
* Psychiatric illness/social situations that would limit consenting and compliance with study requirements.
* Patients with history of hypersensitivity to monoclonal antibodies
* Subjects who are pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raquibul Hannan, MD, PhD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab and SABR
Started | 7
Completed | 2
Not Completed | 5
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
Age, Continuous [Median (Standard Deviation); unit: years] | 57 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3
  Non-White | 4
Region of Enrollment [Number; unit: participants]
  United States | 7
AJCC Stage at Diagnosis [Number; unit: number of participants] — AJCC (American Joint Committee on Cancer ) staging system is a system to describe the amount and spread of cancer in a patient's body, using TNM. T describes the size of the tumor and any spread of cancer into nearby tissue; N describes spread of cancer to nearby lymph nodes; and M describes metastasis (spread of cancer to other parts of the body) by use of x-rays, lab tests, and other tests or procedures.
  Stage 0: Abnormal cells are present but have not spread to nearby tissue; Stage I-III: Cancer is present; Stage IV: The cancer has spread to distant parts of the body.
  number of participants
    Stage III | 4
    Stage IV | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: The primary objective of the randomized phase II trial will be to increase the RR (response rate) of treatment with Nivolumab by the concurrent administration of SAbR. The assessment of RR will be based on the evaluation of ir-RECIST (Response Evaluation Criteria in Solid Tumors) criteria and radiated lesions will be excluded from target lesions. Treatment response will be measured using both the RECIST and immune related RECIST criteria (ir-RECIST), a minor modification of RECIST 1.1 for immunotherapy. Radiated lesions will be excluded from target lesions.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
percentage of participants | 28.6

2. Secondary Outcome: Overall Survival
Description: To evaluate the overall survival (OS), which is defined as the time between date of registration and the date of death due to any cause. In analyzing OS, we will take into account the MSKCC (Memorial Sloan Kettering Cancer Center) prognostic criteria for mRCC (Metastatic Renal Cell Carcinoma) and compare our data to historical controls in the appropriate risk category.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
percentage of participants | 85

3. Secondary Outcome: Progression Free Survival
Description: To evaluate progression free survival (PFS), which is defined as the time between date of registration and the first date of documented disease progression or date of death due to any cause. Progression will be defined according to the ir-RECIST (Response Evaluation Criteria in Solid Tumors) criteria and verified by a second set of imaging at least 6 weeks apart.
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
months | 3.9 [1.9 to 16.5]

4. Secondary Outcome: Complete Response Rate
Description: To evaluate and compare complete response rate in each arm, which is defined as the percentage of patients who show complete response as per ir-RECIST (Response Evaluation Criteria in Solid Tumours) criteria. Treatment response will be measured using both the RECIST and immune related RECIST criteria (ir-RECIST), a minor modification of RECIST 1.1 for immunotherapy. Radiated lesions will be excluded from target lesions.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
Participants | 0

5. Secondary Outcome: Time to Progression
Description: To evaluate and compare time to progression (TTP), which is defined as time between date of registration and date of documented progression, between the experimental and control arms. Progression will be defined according to the ir-RECIST (Response Evaluation Criteria in Solid Tumors) criteria and verified by a second set of imaging at least 6 weeks apart.
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
months | 3.2 [1.8 to 6.3]

6. Secondary Outcome: Median Response Duration
Description: To evaluate median response duration, which is defined as the time between the date of PR (partial response) was first seen until date of progression.
Time Frame: 3 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
weeks | 12 [8.4 to 15.0]

7. Secondary Outcome: Median Response Duration to CR (Complete Response)
Description: To evaluate median duration, which is defined as the time between the date of CR (complete response) was first seen until date of progression.
Time Frame: 3 years
Population: No patient achieved complete response (CR).
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 0

8. Secondary Outcome: Adverse Events
Description: To evaluate the tolerability and toxicity as measured according to CTCAE v4.0. Adverse events will be graded by a numerical score according to the defined NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) and version number 4.0. Adverse events not specifically defined in the NCI CTCAE will be scored on the Adverse Event log according to the general guidelines provided by the NCI CTCAE and as outlined below.
  Grade 1: Mild Grade 2: Moderate Grade 3: Severe or medically significant but not immediately life threatening Grade 4: Life threatening consequences Grade 5: Death related to the adverse event
Time Frame: 3 years
Measure: Number; unit: events
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
events | 58

9. Secondary Outcome: Health-related Quality of Life Using FACT-G Questionnaire (Functional Assessment of Cancer Therapy-General)
Description: FACT-G is a measure that sums the functional well being (FWB), physical well being (PWB), the social/family well-being (S/FWB), and emotional well being (EMB) using a 5-point Likert-type response choices (0 = not at all; 1 = a little bit; 2 =somewhat; 3 = quite a bit; 4 = very much). Questions are phrased so that higher numbers indicate a better health state, leading to some items being reverse-scored. Scoring the FACT-G is performed through a simple sum of item scores with a total possible score of 105.
Time Frame: Baseline and 6 months
Measure: Median (Full Range); unit: score on scale
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
score on scale
  Baseline | 70.933 [29 to 103]
  6 month follow up | 79 [29 to 96]

10. Secondary Outcome: Health-related Quality of Life Using EQ-5D (European Quality of Life Five Dimension) Questionnaire With VAS (Visual Analogue Scale)
Description: EQ-5D is a standardized participant completed questionnaire consisted of 2 components: a health state profile and VAS. EQ-5D health state profile had 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Responses to 5 dimensions comprised a health state/a single utility index value. Every health state (coded as combination of responses on each of 5 dimensions) had a unique predefined utility index value assigned to it, by EuroQol. US value sets (with all possible health states) was used for adults in the study, range from 1 to -0.109. Higher (positive) scores = better health state. VAS was used to record a participant's rating for his/her current health-related quality of life state and captured on a vertical VAS (0-100), where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline and 6 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
score on a scale
  Baseline Mobility | 1 [1 to 5]
  6 month follow up Mobility | 1 [1 to 5]
  Baseline Self-Care | 1 [1 to 5]
  6 month follow up Self-Care | 1 [1 to 5]
  Baseline Usual Activities | 1 [1 to 5]
  6 month follow up Usual Activities | 4 [1 to 5]
  Baseline Pain/Discomfort | 2 [1 to 5]
  6 month follow up Pain/Discomfort | 3 [1 to 5]
  Baseline Anxiety/Depression | 1 [1 to 5]
  6 month follow up Anxiety/Depression | 1 [1 to 5]
  Baseline EQ-VAS | 90 [1 to 100]
  6 month follow up EQ-VAS | 90 [1 to 100]

11. Secondary Outcome: Health-related Quality of Life Using FKSI (Functional Assessment of Cancer Therapy-Kidney Symptom Index) Questionnaire
Description: The FKSI is a 15 question validated symptom index for kidney cancer patients. This scale focuses on symptoms predominantly related to kidney cancer such as energy, fatigue, pain, bone pain, weight loss, shortness of breath, cough, fever, hematuria. Each item was scored on a 5-point scale (0=not at all to 4=very much). FKSI total score ranged from 0 (most severe symptoms) to 60 (no symptoms) with a higher score indicating a better outcome.
Time Frame: Baseline and 6 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Nivolumab and SABR
Number analyzed (Participants) | 7
score on a scale
  Baseline | 46 [31 to 55]
  6 month follow up | 48 [24 to 50]

12. Other Pre Specified Outcome: Immunological Biomarkers
Description: To identify immunological biomarkers as predictors of treatment response or resistance. This is an exploratory outcome and was added as a secondary outcome in error.
Time Frame: 3 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Cost-effectiveness
Description: To evaluate the cost-effectiveness and cost-utility of the addition of SAbR to Nivolumab in patients with mRCC. This is an exploratory outcome and was added as a secondary outcome in error.
Time Frame: 3 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Immunogenicity
Description: To measure and compare treatment-related tumor-specific immune response (immunogenicity) in each arm. This is an exploratory outcome and was added as a secondary outcome in error.
Time Frame: 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse events will be graded by a numerical score according to the defined NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening; Grade 4: Life threatening consequences; Grade 5: Death related to the adverse event
Arm/Group | Nivolumab and SABR
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and SABR (N=7)
Gastrointestinal (Gastrointestinal disorders) | 7 (25)
Genitourinary (Renal and urinary disorders) | 2 (2)
Hematologic (Blood and lymphatic system disorders) | 7 (7)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 (5)
Renal/Electrolyte (Renal and urinary disorders) | 2 (2)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Skin (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT02781506/Prot_SAP_000.pdf